CLINICAL TRIAL: NCT07199465
Title: A Phase 1, Open-label, Single-arm Study to Evaluate the Pharmacokinetics and Safety of Letermovir in Pediatric Kidney Transplant (KT) Recipients Less Than 18 Years of Age and Weighing Less Than 40 Kilograms
Brief Title: A Clinical Study of Letermovir (MK-8228) in Children and Adolescents Who Receive a Kidney Transplant (KT) (MK-8228-077)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8228-077; MK-8228-077 (Other: MSD)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Cytomegalovirus Prophylaxis
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Weight-banded letermovir dosing (Experimental): Participants who are between 4 and 52 weeks post-KT will receive letermovir for 7 consecutive days.
  Interventions: Drug: Letermovir

INTERVENTIONS:
Drug: Letermovir — Administered orally (as tablets/pellets) or via gastrostomy or nasogastric tube (as pellets) for 7 consecutive days.
  Other Names: MK-8228; AIC246; AIC001; PREVYMIS™

SUMMARY:
Researchers are looking for a way to prevent cytomegalovirus (CMV) in children and adolescents who receive a kidney transplant (KT) and weigh less than 40 kilograms (88.2 pounds). The goals of the study are to:

* Learn what happens to letermovir in the body over time
* Learn about the safety of letermovir and if participants tolerate it

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is a recipient of a primary or secondary allograft kidney
* Is at least 4 weeks posttransplant and not more than 52 weeks posttransplant at the time of enrollment (Day 1) and is being managed per local standard of care
* Has stable kidney function posttransplant
* Has undetectable CMV deoxyribonucleic acid (DNA) from a plasma or whole blood sample collected within 14 days prior to enrollment
* Must be able to take (as assessed by the investigator) letermovir tablets or oral pellets by mouth, or via gastrostomy or nasogastric tube (oral pellets only)
* Does not have a condition that may interfere with the absorption of oral medication (e.g., vomiting, diarrhea, or a malabsorptive condition) from the day of enrollment (Day 1) until the intensive pharmacokinetics (IPK) sampling is completed
* Weighs ≥2.5 and <40 kg at enrollment (Day 1)

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has CMV disease or suspected CMV disease between screening and enrollment
* Is on dialysis or plasmapheresis at the time of enrollment
* Has evidence of CMV viremia at any time from screening until the time of enrollment
* Has Child-Pugh B or C hepatic insufficiency within 14 days before enrollment
* Is a multi-organ transplant recipient (e.g., kidney-pancreas)
* Has any uncontrolled infection on the day of enrollment
* Requires mechanical ventilation, or is hemodynamically unstable, at the time of enrollment
* Has received or is receiving protocol-specified prohibited medications

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2028-04-14 (Estimated); Study Completion 2028-05-19 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve From Time 0 to 24 Hours (AUC0-24) | Day 7: Predose and at designated timepoints post-dose (up to 24 hours)
  Blood samples will be collected at multiple time points to estimate AUC0-24

SECONDARY OUTCOMES:
Percentage of Participants Who Experience an Adverse Event (AE) | Up to 21 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experienced an AE is reported.
Percentage of Participants Who Discontinue Study Intervention Due to an AE | Up to 7 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinued study treatment due to an AE is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- United States (6):
  - Lucile Packard Children's Hospital ( Site 0001), Palo Alto, California
  - University of Michigan ( Site 0014), Ann Arbor, Michigan
  - Mayo Clinic - Rochester ( Site 0015), Rochester, Minnesota
  - Morgan Stanley Children's Hospital ( Site 0018), New York, New York
  - Duke University Medical Center ( Site 0008), Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center ( Site 0002), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com